CLINICAL TRIAL: NCT01570686
Title: An 8-week Randomized, Open-label, Multi-center Study to Evaluate the Efficacy and Safety of Oral Aliskiren 300 mg Once Daily Under Light Meal Versus Fasted Condition in Patients With Hypertension
Brief Title: 8-week Randomized, Open-label Study to Evaluate Food Effect on Efficacy and Safety of Oral Aliskiren 300 mg in Patients With Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPP100A2413; 2011-005297-36 (EudraCT Number)
Record Dates: First submitted 2012-04-02; First posted 2012-04-04 (Estimated); Results first posted 2014-01-01 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Hypertension
Keywords: Food effect, hypertension, aliskiren
MeSH Terms: conditions — Hypertension | interventions — aliskiren

ARMS (2):
- Aliskiren: Fed (Experimental): Aliskiren 300 mg once daily, taken 30 minutes after start of light breakfast
  Interventions: Drug: Aliskiren
- Aliskiren: Fasting (Experimental): Aliskiren 300 mg once daily taken after after an overnight fast
  Interventions: Drug: Aliskiren

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 300 mg once daily
  Other Names: Tekturna, rasilez

SUMMARY:
The purpose of this study is to evaluate the effect of food on aliskiren's efficacy, pharmacokinetics and safety following an oral dose of 300 mg, given once daily under light meal versus fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with essential hypertension, untreated or currently taking antihypertensive therapy (monotherapy or combination therapy).
* Patients with an office BP ≥ 140/90 mmHg and < 180/110mmHg at the randomization visit and the preceding visit
* Patients must have an absolute difference of ≤ 10 mmHg in both their msSBP and their msDBP between the randomization visit and the preceding visit

Exclusion Criteria:

* Malignant hypertension or severe hypertension (grade 3 of WHO classification; msSBP ≥180 mmHg or msDBP ≥110 mmHg)
* History or evidence of a secondary form of hypertension, such as renal parenchymal hypertension, renovascular hypertension, coarctation of the aorta, primary hyperaldosteronism, Cushing's disease, drug-induced hypertension, unilateral or bilateral renal artery stenosis, pheochromocytoma, polycystic kidney disease (PKD).
* Type 1 or Type 2 diabetes mellitus with a fasting glycosylated hemoglobin (HbA1c) > 8%
* Evidence of renal impairment as determined by one of the following: serum creatinine >1.5 x ULN or eGFR < 30 ml/min/1.73m2 at Visit 1, a history of dialysis, or a history of nephrotic syndrome

Other protocol-defined inclusion/exclusion criteria may apply.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 589 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (79):
- United States (41):
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, Walnut Creek, California
  - Novartis Investigative Site, Westlake Village, California
  - Novartis Investigative Site, Coral Gables, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, South Miami, Florida
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Opelousas, Louisiana
  - Novartis Investigative Site, Chaska, Minnesota
  - Novartis Investigative Site, Edina, Minnesota
  - Novartis Investigative Site, Saint Paul, Minnesota
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Picayune, Mississippi
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Salisbury, North Carolina
  - Novartis Investigative Site, Shelby, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Lyndhurst, Ohio
  - Novartis Investigative Site, Marion, Ohio
  - Novartis Investigative Site, Norman, Oklahoma
  - Novartis Investigative Site, Eugene, Oregon
  - Novartis Investigative Site, Oregon City, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Beaumont, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Lake Jackson, Texas
  - Novartis Investigative Site, Pasadena, Texas
  - Novartis Investigative Site, Centerville, Utah
  - Novartis Investigative Site, Arlington, Virginia
  - Novartis Investigative Site, Ettrick, Virginia
  - Novartis Investigative Site, Midlothian, Virginia
  - Novartis Investigative Site, Port Orchard, Washington
- Canada (6):
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Mirabel, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
- Italy (3):
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Sassari, SS
- Puerto Rico (3):
  - Novartis Investigative Site, Carolina
  - Novartis Investigative Site, Cidra
  - Novartis Investigative Site, Manatí
- Slovakia (14):
  - Novartis Investigative Site, Banská Bystrica, Slovak Republic
  - Novartis Investigative Site, Bratislava, Slovak Republic
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Nitra, Slovak Republic
  - Novartis Investigative Site, Rimavská Sobota, Slovak Republic
  - Novartis Investigative Site, Senec, Slovak Republic
  - Novartis Investigative Site, Snina, Slovak Republic
  - Novartis Investigative Site, Svidník, Slovak Republic
  - Novartis Investigative Site, Trnava, Slovak Republic
  - Novartis Investigative Site, Bratislava, Slovakia
  - Novartis Investigative Site, Martin, Slovakia
  - Novartis Investigative Site, Prešov, Slovakia
  - Novartis Investigative Site, Šaľa, Slovakia
  - Novartis Investigative Site, Zvolen, Slovakia
- Spain (8):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Centelles, Catalonia
  - Novartis Investigative Site, Corbera de Llobregat, Catalonia
  - Novartis Investigative Site, Hostalets de Balenya, Catalonia
  - Novartis Investigative Site, Vic, Catalonia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Alzira, Valencia
  - Novartis Investigative Site, Quart de Poblet, Valencia
- Taiwan (4):
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan, ROC
  - Novartis Investigative Site, Changhua

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 691 patients enrolled in the study with 590 patients randomized. 1 patient was mis-randomized and did not receive study medication, therefore 589 patients actually received study medication.
Period: Overall Study
Arm/Group | Aliskiren: Fed | Aliskiren: Fasting
Started | 296 | 294
Safety and Full Analysis Set (FAS) | 295 (One patient was mis-randomized and never received study drug. Hence not included in Safety or FAS.) | 294
Completed | 274 | 278
Not Completed | 22 | 16
Not completed — Abnormal test procedure result(s) | 1 | 1
Not completed — Administrative problems | 0 | 1
Not completed — Adverse Event | 8 | 6
Not completed — Lost to Follow-up | 4 | 3
Not completed — Protocol Deviation | 3 | 0
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Unsatisfactory therapeutic effect | 2 | 1

BASELINE CHARACTERISTICS:
Population: All Randomized patients (including one mis-randomized patient in Aliskiren:Fed arm).
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren: Fed | Aliskiren: Fasting | Total
Number analyzed (Participants) | 296 | 294 | 590
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.7 (10.44) | 56.1 (11.03) | 55.9 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 126 | 278
  Male | 144 | 168 | 312

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Visit 3) to End of Study (Week 8) in Mean 24 Hour Ambulatory Systolic Blood Pressure (maSBP)
Description: 24 hour ambulatory blood pressure measurement (ABPM) were taken twice, at baseline and at the end of 8 weeks. An Ambulatory Blood Pressure Monitoring device (ABPM) was attached to the non-dominant arm. The mean change of 24 hours maSBP from baseline to week 8 was estimated using an Analysis of Covariance (ANCOVA) model by using treatment, region as factors, and baseline as covariate.
Time Frame: Baseline, week 8
Population: Full Analysis Set (FAS): consisted of all randomized patients. Mis-randomized patients were excluded from the FAS. Patients with ABPM measurements at both baseline and week 8 were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren: Fed | Aliskiren: Fasting
Number analyzed (Participants) | 263 | 266
mmHg | -7.03 (0.50) | -7.79 (0.50)

2. Secondary Outcome: Change From Baseline (Visit 3) to End of Study (Week 8) in Mean 24 Hour Ambulatory Diastolic Blood Pressure (maDBP)
Description: 24 hour ambulatory blood pressure measurement (ABPM) were taken twice, at baseline and at the end of 8 weeks. An Ambulatory Blood Pressure Monitoring device (ABPM) was attached to the non-dominant arm. The mean change of 24 hours maDBP from baseline to week 8 was estimated using an Analysis of Covariance (ANCOVA) model by using treatment, region as factors, and baseline as covariate.
Time Frame: Baseline, week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren: Fed | Aliskiren: Fasting
Number analyzed (Participants) | 263 | 266
mmHg | -4.01 (0.31) | -4.39 (0.31)

3. Secondary Outcome: Percentage of Patients Achieving Blood Pressure Control
Description: Patients achieving blood pressure control were patients who, at week 8, had a mean sitting systolic blood pressure (msSBP)/ mean sitting diastolic blood pressure (msDBP) < 140/90 mmHg
Time Frame: 8 weeks
Population: Full Analysis Set (FAS): consisted of all randomized patients. Mis-randomized patients were excluded from the FAS. Patients with mean sitting blood pressure measurement over 8 weeks were included in this analysis.
Measure: Number; unit: Percentage of patients
Arm/Group | Aliskiren: Fed | Aliskiren: Fasting
Number analyzed (Participants) | 293 | 294
Percentage of patients | 44.7 | 41.5

4. Secondary Outcome: Change From Baseline (Visit 3) to End of Study (8 Weeks) in Mean Sitting Systolic Blood Pressure (msSBP) and Mean Sitting Diastolic Blood Pressure (msDBP)
Description: Sitting blood pressure (BP) was measured at trough (approximately 24 hours ± 3 hours post dose) and recorded at all study visits. At the first study visit, the BP was checked in both arms and the arm with higher systolic BP (SBP) was used for all subsequent readings throughout the study. At each study visit, after the patient had been sitting for five minutes, systolic and diastolic blood pressures (msSBP and msDBP) were measured four times using a standard mercury sphygmomanometer and appropriate size cuff. The repeat sitting measurements were made at 2 minute intervals and the mean of all four sitting blood pressure measurements was used as the average sitting office blood pressure for that visit. The analysis of covariance (ANCOVA) model used treatment, region as factors, and baseline as covariate.
Time Frame: Baseline, Week 8
Population: Full Analysis Set (FAS): consisted of all randomized patients. Mis-randomized patients were excluded from the FAS. Patients with official mean sitting blood pressure measurements both at baseline and week 8 were icluded in this analysis.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren: Fed | Aliskiren: Fasting
Number analyzed (Participants) | 293 | 294
mmHg
  Mean sitting SBP (msSBP) | -13.65 (0.85) | -13.98 (0.85)
  Mean sitting DBP (msDBP) | -8.97 (0.50) | -8.56 (0.50)

5. Secondary Outcome: Percentage of Patients Achieving a Successful Response in Systolic Blood Pressure Reduction
Description: Successful response in systolic blood pressure reduction at end of 8-week treatment was defined as msSBP <140 mmHg or a reduction in msSBP ≥ 20 mmHg from baseline.
Time Frame: Baseline, Week 8
Population: Full Analysis Set (FAS): consisted of all randomized patients. Mis-randomized patients were excluded from the FAS. Patients with mean sitting SBP measurement at baseline and over 8 weeks were included in this analysis.
Measure: Number; unit: Percentage of patients
Arm/Group | Aliskiren: Fed | Aliskiren: Fasting
Number analyzed (Participants) | 293 | 294
Percentage of patients | 54.9 | 55.8

6. Secondary Outcome: Pharmacokinetic (PK) of Aliskiren: The Observed Maximum Plasma Concentration (Cmax) Following Drug Administration in Fasted vs. Fed
Description: Blood samples were collected at Week 4 and Week 8 in a subset of patients (approximately 15% of each treatment group) for PK analysis.
Time Frame: Week 4 (0, 0.5, 1, 1.5, 2, 4, 6 and 24 hrs post-dose) and week 8 (0, 0.5, 1, 1.5, 2, 4, 6 and 24 hrs post-dose)
Population: Pharmacokinetics set included all patients who had evaluable aliskiren concentration data with no protocol deviations that presumably affect PK results were included in the pharmacokinetic evaluations
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Aliskiren: Fed | Aliskiren: Fasting
Number analyzed (Participants) | 46 | 53
ng/mL
  Week 4 (Day 28) (N= 46, 52) | 108 (153) | 273 (276)
  Week 8 (Day 56) (N= 42, 53) | 102 (139) | 252 (220)

7. Secondary Outcome: Pharmacokinetic of Aliskiren: The Area Under the Plasma Concentration-time Curve From Time Zero to the End of the Dosing Interval Tau (AUCtau) in Fasted vs. Fed
Description: as for outcome 6
Time Frame: Week 4 (0, 0.5, 1, 1.5, 2, 4, 6 and 24 hrs post-dose) and week 8 (0, 0.5, 1, 1.5, 2, 4, 6 and 24 hrs post-dose)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Aliskiren: Fed | Aliskiren: Fasting
Number analyzed (Participants) | 46 | 53
ng*h/mL
  Week 4 (Day 28) (N= 44, 50) | 872 (603) | 1580 (1120)
  Week 8 (Day 56) (N= 40, 51) | 1100 (1620) | 1540 (1120)

8. Secondary Outcome: Pharmacokinetic of Aliskiren: Time to Reach the Maximum Concentration (Tmax) After Drug Administration in Fasted vs. Fed
Description: as for outcome 6
Time Frame: Week 4 (0, 0.5, 1, 1.5, 2, 4, 6 and 24 hrs post-dose) and week 8 (0, 0.5, 1, 1.5, 2, 4, 6 and 24 hrs post-dose)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Aliskiren: Fed | Aliskiren: Fasting
Number analyzed (Participants) | 46 | 53
Hour
  Week 4 (Day 28) (N=46, 52) | 2.60 (1.68) | 1.71 (1.45)
  Week 8 (Day 56) (N= 42, 53) | 3.33 (3.71) | 1.72 (3.32)

9. Secondary Outcome: Change From Baseline to Week 8 in Plasma Renin Activity (PRA)
Description: Biomarkers related to hypertension-related pathophysiology were evaluated in this study, such as plasma renin activity (PRA) . Blood samples were taken at Visit 3 (baseline) and Visit 6 (week 8).The difference between baseline and week 8 was calculated.
Time Frame: Baseline, Week 8
Population: Full Analysis Set (FAS): consisted of all randomized patients. Mis-randomized patients were excluded from the FAS. Patients with both baseline and week 8 measurement for PRA are included in this analysis.
Measure: Mean (Standard Deviation); unit: ng/mL/hr
Arm/Group | Aliskiren: Fed | Aliskiren: Fasting
Number analyzed (Participants) | 42 | 47
ng/mL/hr | -0.519 (1.4016) | -1.962 (6.7419)

10. Secondary Outcome: Change From Baseline to Week 8 in Plasma Renin Concentration (PRC)
Description: Biomarkers related to hypertension-related pathophysiology were evaluated in this study, such as plasma renin concentration (PRC). Blood samples were taken at Visit 3 (baseline) and Visit 6 (week 8). The difference between baseline and week 8 was calculated.
Time Frame: Baseline, Week 8
Population: Full Analysis Set (FAS): consisted of all randomized patients. Mis-randomized patients were excluded from the FAS. Patients with both baseline and week 8 measurement for PRC are included in this analysis.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Aliskiren: Fed | Aliskiren: Fasting
Number analyzed (Participants) | 42 | 47
ng/L | 37.881 (63.4412) | 50.967 (81.8987)

11. Secondary Outcome: Number of Patients With Adverse Events, Serious Adverse Events and Death
Time Frame: 8 weeks
Population: Safety Set (SAF): consisted of all patients who received at least one dose of randomized study medication.
Measure: Number; unit: Patients
Arm/Group | Aliskiren: Fed | Aliskiren: Fasting
Number analyzed (Participants) | 295 | 294
Patients
  Any Adverse event | 73 | 90
  Serious Adverse events | 4 | 2
  Death | 0 | 0

ADVERSE EVENTS:
Description: Safety Set (SAF): consisted of all patients who received at least one dose of randomized study medication.
Groups:
- Aliskiren 300 mg (Fasted): Aliskiren 300 mg once daily taken after after an overnight fast
Arm/Group | Aliskiren: Fed | Aliskiren 300 mg (Fasted)
Serious Adverse Events (participants affected / at risk) | 4/295 | 2/294
Other Adverse Events (participants affected / at risk) | 3/295 | 16/294
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren: Fed (N=295) | Aliskiren 300 mg (Fasted) (N=294)
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren: Fed (N=295) | Aliskiren 300 mg (Fasted) (N=294)
Diarrhoea (Gastrointestinal disorders) | 3 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.